CLINICAL TRIAL: NCT02793869
Title: A Novel Congenital Cataract Category System Based on Lens Opacity Positions and Their Relevant Anterior Segment Characteristics
Brief Title: A Novel Congenital Cataract Category System
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: CCPMOH2016-China-4
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Cataract
Keywords: congenital cataract;anterior segment characteristics
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Total cataract group: All selected eyes were categorized into four groups: total cataracts, anterior cataracts, interior cataracts and posterior cataracts, based on the position of lens opacities shown by both a slit lamp (BX900, HAAG-STREIT AG, Bern, Switzerland) examination and a 3-dimensional anterior segment imaging and analysis system (Pentacam HR, Oculus Inc., Wetzlar, Germany) after mydriasis.
- Anterior cataract group: All selected eyes were categorized into four groups: total cataracts, anterior cataracts, interior cataracts and posterior cataracts, based on the position of lens opacities shown by both a slit lamp (BX900, HAAG-STREIT AG, Bern, Switzerland) examination and a 3-dimensional anterior segment imaging and analysis system (Pentacam HR, Oculus Inc., Wetzlar, Germany) after mydriasis.
- Interior cataracts group: All selected eyes were categorized into four groups: total cataracts, anterior cataracts, interior cataracts and posterior cataracts, based on the position of lens opacities shown by both a slit lamp (BX900, HAAG-STREIT AG, Bern, Switzerland) examination and a 3-dimensional anterior segment imaging and analysis system (Pentacam HR, Oculus Inc., Wetzlar, Germany) after mydriasis.
- Posterior cataract group: All selected eyes were categorized into four groups: total cataracts, anterior cataracts, interior cataracts and posterior cataracts, based on the position of lens opacities shown by both a slit lamp (BX900, HAAG-STREIT AG, Bern, Switzerland) examination and a 3-dimensional anterior segment imaging and analysis system (Pentacam HR, Oculus Inc., Wetzlar, Germany) after mydriasis.

SUMMARY:
Congenital cataracts (CC) are the leading cause of childhood visual disabilities and treatable childhood blindness worldwide1. CC patients have a wide range of presentations of lens opacities and are generally categorized into several groups based on the etiologies, anatomical positions, or shapes of lens opacities. Cataractous eyes of CC patients are also frequently complicated with other anterior segment abnormalities due to their close anatomical relationships and similar developmental origins. Lens opacities in different positions may be related to specific anterior segment abnormalities; for example, anterior polar cataracts are associated with greater corneal astigmatism (CA). However, no studies have systematically related the position of lens opacities to specific anterior segment abnormities, mainly due to the small number of CC patients, a lack of proper equipment, and a lack of awareness of these important relationships.

DETAILED DESCRIPTION:
Congenital cataracts (CC) are the leading cause of childhood visual disabilities and treatable childhood blindness worldwide1. CC patients have a wide range of presentations of lens opacities and are generally categorized into several groups based on the etiologies, anatomical positions, or shapes of lens opacities. Cataractous eyes of CC patients are also frequently complicated with other anterior segment abnormalities due to their close anatomical relationships and similar developmental origins. Lens opacities in different positions may be related to specific anterior segment abnormalities; for example, anterior polar cataracts are associated with greater corneal astigmatism (CA). However, no studies have systematically related the position of lens opacities to specific anterior segment abnormities, mainly due to the small number of CC patients, a lack of proper equipment, and a lack of awareness of these important relationships.

Using the largest CC database in the Zhongshan Ophthalmic Center (ZOC), the current study compared the anterior segment characteristics of CC patients with lens opacities in different positions and further proposed a modified CC category system based on the specific relationships between the position of lens opacities and anterior segment characteristics. Knowledge of these relationships is beneficial for further understanding of CC occurrence and development and has clinical significance for CC diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital cataract
* less than 18 years old

Exclusion Criteria:

* With other ocular abnormalities including severe corneal diseases, lens luxation, glaucoma, retinal diseases, nystagmus, nanophthalmos, and strabismus.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This was a prospective study and was included in our series of ongoing studies at the Childhood Cataract Program of the Chinese Ministry of Health (CCPMOH), a national project for congenital cataract (CC) treatment and research. CC patients less than 18 years old and seeking treatment at the ZOC, one of the best eye care facilities in China, from February 2011 to December 2015 were candidates for this study. All included participants were diagnosed with CC before surgery and lacked other ocular abnormalities, such as severe corneal diseases, lens luxation, glaucoma, retinal diseases, nystagmus, nanophthalmos, and strabismus. A total of 428 CC patients were included.
Sampling Method: Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2011-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The mean keratometry value | Baseline
  The anterior segment parametersthe mean keratometry value of CC patients were measured by the 3-dimensional anterior segment imaging analysis system.
The central corneal thickness | Baseline
  The anterior segment parametersthe central corneal thickness of CC patients were measured by the 3-dimensional anterior segment imaging analysis system.
The anterior chamber depth | Baseline
  The anterior segment parametersthe anterior chamber depth of CC patients were measured by the 3-dimensional anterior segment imaging analysis system.

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D., Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Weirong Chen, M.D., Ph.D, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lin H, Long E, Chen W, Liu Y. Documenting rare disease data in China. Science. 2015 Sep 4;349(6252):1064. doi: 10.1126/science.349.6252.1064-b. No abstract available. PMID 26339020
- See also: Description Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/
- See also: Homepage of Childhood Cataract Program of the Chinese Ministry of Health(CCPMOH) — http://www.cnccclub.com/